CLINICAL TRIAL: NCT01285141
Title: Phase I Clinical Trial in Healthy Female Volunteers of Reactogenicity and Immunogenicity of Three Cervico-vaginal Topical Immunisations With a Fixed Dose of HIV CN54gp140 Glycoprotein-hsp70 Conjugate Vaccine
Brief Title: Reactogenicity and Immunogenicity of Cervico-vaginal CN54gp140-hsp70 Conjugate Vaccine
Acronym: TL01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, David JM Lewis, Professor of Clinical Vaccinology, St George's, University of London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010-022740-20
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: HIV Infections
Keywords: HIV Infections; Acquired Immune Deficiency Syndrome
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaginal immunisation (Experimental): CN54gp140 glycoprotein-hsp70 conjugate vaccine
  Interventions: Biological: CN54gp140 glycoprotein-hsp70 conjugate vaccine

INTERVENTIONS:
Biological: CN54gp140 glycoprotein-hsp70 conjugate vaccine — CN54gp140-hsp70 conjugate vaccine administered intravaginally 3 times over a 12-week period
  Other Names: ZM96gp140 glycoprotein

SUMMARY:
A vaccine to prevent infection with the Human Immunodeficiency Virus (HIV) is urgently needed. Worldwide, most HIV infections occur through sex between a man and woman. The vaccine in this study consists of a protein from HIV that has been synthetically produced and linked to a protein that boosts immune responses. It has not been tested in humans before, but it is expected (from animal studies) that direct application into the female genital tract (via the vagina) as liquid drops, will provoke immune protection at the site of HIV infection. This is less applicable to men, therefore only healthy, HIV negative women will be recruited. The investigators will recruit at one site, which is a university vaccine research centre with experience of running similar trials. The study will last 24 weeks during which subjects will have blood samples taken on six visits, and three immunisations over 12 weeks in which 1 millilitres of vaccine is placed into the vaginal by inserting a small plastic syringe. The purpose of this initial small study is to monitor safety of the vaccine and to determine whether it is appropriate to continue into future, larger studies in which the immune response to the vaccine is measured.

DETAILED DESCRIPTION:
This hypothesis-generating, first-in-human, Phase 1 study will be conducted according to the Standard Operating Procedures (SOPs) of St George's. The purpose of the study is to determine the immediate safety and reactogenicity of the vaccine, to guide future larger Phase 1/2 studies of safety and efficacy.

Eight subjects will be included to receive 3 cervico-vaginal topical applications of 100µg of CN54gp140-hsp70 conjugate vaccine in 1.0 mL physiological buffer, administered as topical intra-vaginal drops on day 0, and at 4 and 12 weeks after the first immunisation. The study will consist of 1 pre-study screening visit, 3 immunisation visits, and 2 follow-up visits over a total period of 20 weeks. Subjects will be recruited as one cohort in two groups of four. The dose of antigens and immunisation schedule has been selected based on pre-clinical and clinical experience with the same HIV envelope protein.

Each subject's medical history (including past and present illnesses, current medications, family medical history) will be formally assessed and recorded at screening. Volunteers' age, gender, height, weight and ethnic origin will be recorded. A full physical examination will be conducted by a registered medical practitioner at screening and the final study visit. Regular assessments of vital signs (pulse, blood pressure, temperature) will be made on all visits.

Diary cards, investigator-prompted recall of events, laboratory tests (haematology, biochemistry) and direct visualisation of immunisation site will be used to identify Adverse Events. Frequency of vaccine-related Adverse Events is the Primary Study Endpoint.

Before and after each immunisation visit (0, 4 and 12 weeks) blood samples will be obtained for collection of serum and for separation of PBMCs for cellular assays. At each time point, vaginal and cervical secretions will be taken. All immunology assays are exploratory and are not study endpoints. HIV serology and DNA detection will be repeated at the final visit to detect subjects who may have contracted HIV infection during the study period, and who may therefore have developed antibody and T-cell responses due to the HIV infection that would interfere with exploratory immunology assays.

ELIGIBILITY:
Inclusion Criteria:

* Adult female volunteers, 18 to 45 years of age, who have signed an informed consent form following a detailed written explanation of participation in the protocol.
* Volunteers who are in good health as determined by medical history, physical examination and clinical judgement.
* Available for the duration of the study.
* Women who, if capable of becoming pregnant during the study, have agreed to have a pregnancy test immediately before immunisation, and to use appropriate contraception methods during the whole study period. Appropriate contraception shall include physician-prescribed oral hormonal agents, barrier contraceptives, regular and consistent use of condoms without spermicidal agents, or intrauterine devices only.
* Agree not to undertake any vaginal practices other than receptive intercourse with a male or use of sanitary tampons during menses. Use of condoms without spermicidal agents is encouraged.
* Have not donated blood during 3 months prior to study entry and agree to not donate for 3 months after the end of their participation in the study

Exclusion Criteria:

* They have hypersensitivity to any component of the vaccine used in this study.
* They are found to be HIV antibody or HIV proviral DNA positive at the time of initial screening.
* They have a known or suspected history of cervico-vaginal disease, malignancy or abnormality discovered at time of screening, or who have undergone a Letts procedure.
* They present in the samples obtained at the screening visit:
* a clinically significant abnormality in the haematological or biochemical assays.
* Positive tests for Hepatitis B and/or C infection
* Positive tests for genital infections: Chlamydia trachomatis, Neisseria gonorrhoea, Treponema pallidum (syphilis).
* An abnormal value will be defined by the ranges quoted by pathology laboratory.
* They have a known or suspected impairment of lung, heart, liver, kidney, blood disorders or immune dysfunction.
* They are receiving immunosuppressive therapy (including systemic steroids).
* They are receiving any regular medications via vaginal route.
* They have any acute infections (including fever greater than or equal to 38°C) or any chronic disease.
* They present a current problem with substance abuse or with a history of substance abuse, which, in the opinion of the investigator, might interfere with participation in the study.
* They have any condition that, in the opinion of the investigator, might interfere with the evaluation of the study objectives.
* They have received an investigational agent within 3 months prior to study entry.
* They cannot speak fluent English
* They are planning to leave the area of the study site prior to the end of the study period, or are likely not to complete the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Frequency of local immunisation site vaccine-related Adverse Events | 20 weeks
  Semi-structured diary card of solicited local symptoms (vaginal irritation, discharge, bleeding), investigator-prompted recall of unsolicited symptoms, recorded for 20 weeks from day of first immunisation. Visual inspection of cervix-vagina by trained operator prior to immunisation and on final visit.

SECONDARY OUTCOMES:
Frequency of generalised vaccine-related Adverse Events | 20
  Semi-structured diary card of solicited generalised symptoms (headache, fever, malaise, chills, myalgia), investigator-prompted recall of unsolicited symptoms, recorded for 20 weeks from day of first immunisation.
Frequency of vaccine-related Adverse Events in hematology and serum biochemistry parameters | 20
  Adverse Events defined as deviation from normal ranges defined for pre-determined panels of hematology and serum biochemistry parameters.
Frequency of subjects mounting a cervico-vaginal antibody response to CN54gp140 | 20 weeks
  Exploratory assay of cervico-vaginal antibody to CN54gp140, measured at each scheduled study visit. Not a study endpoint.
Frequency of subjects mounting a cervico-vaginal antibody response to hsp70 | 20 weeks
  Exploratory assay of cervico-vaginal antibody to hsp70, measured at each scheduled study visit. Not a study endpoint.
Frequency of subjects mounting a T cellular proliferative response to CN54gp140 | 20 weeks
  Exploratory assay of T cell proliferation in response to in vitro antigen stimulation, measured at each scheduled study visit. Not a study endpoint.
Frequency of subjects mounting a serum antibody response to CN54gp140 | 20 weeks
  Exploratory assay of serum antibody to CN54gp140, measured at each scheduled study visit. Not a study endpoint.
Frequency of subjects mounting a serum antibody response to hsp70 | 20 weeks
  Exploratory assay of serum antibody to hsp70, measured at each scheduled study visit. Not a study endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: David JM Lewis, MD, Principal Investigator — St George's, University of London, UK
Locations (1):
- St George's - University of London, London, England, United Kingdom

REFERENCES:
- [Derived] Lewis DJ, Wang Y, Huo Z, Giemza R, Babaahmady K, Rahman D, Shattock RJ, Singh M, Lehner T. Effect of vaginal immunization with HIVgp140 and HSP70 on HIV-1 replication and innate and T cell adaptive immunity in women. J Virol. 2014 Oct;88(20):11648-57. doi: 10.1128/JVI.01621-14. Epub 2014 Jul 9. PMID 25008917
- See also: St George's, University of London — http://www.sgul.ac.uk